CLINICAL TRIAL: NCT05618899
Title: Effect oh High Intensity Interval Training Versus Moderate Intensity Exercises on Physical Health and Cardiorespiratory Fitness in Obeses Women
Brief Title: Effect of Exercises on Physical Health and Cardiorespiratory Fitness in Obese Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/22/0343 MAHAM ATHAR
Record Dates: First submitted 2022-11-08; First posted 2022-11-16 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Obesity
Keywords: High intensity exercise; Moderate intensity exercise
MeSH Terms: conditions — Obesity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIGH INTENSITY INTERVAL TRAINING (Experimental): High intensity interval training basicaaly short bursts of intense exercise alternating with low intensity recovery periods. Training should be done on treadmill for 25-30 minutes.. Training proceed for 1 month once a day
  Interventions: Other: HIGH INTENSITY INTERVAL TRAINING
- MODERATE INTENSITY EXERCISE (Experimental): moderate intensity exercises consist of generally 30-60 minutes of aerobic exercises at 64-76% of peak heart rate. Training should be done on treadmill for 30-60 minutes. Training proceed for 1 month once a day
  Interventions: Other: MODERATE INTENSITY EXERCISE

INTERVENTIONS:
Other: HIGH INTENSITY INTERVAL TRAINING — Training should be done on treadmill for 25-30 minutes.. Training proceed for 1 month once a day
  Arms: HIGH INTENSITY INTERVAL TRAINING
Other: MODERATE INTENSITY EXERCISE — moderate intensity exercises consist of generally 30-60 minutes of aerobic exercises at 64-76% of peak heart rate. Training should be done on treadmill for 30-60 minutes. Training proceed for 1 month once a day
  Arms: MODERATE INTENSITY EXERCISE

SUMMARY:
The study will be a Randomized clinical trial and will be conducted in services hospital lahore. The sample size of 50 patients will be taken in this study to find the effects of high intensity interval training versus moderate intensity exercises on physical health and cardiorespiratory fitness in obese women.

Patients will be divided into two groups (Group A will be treated with high intensity interval training and Group B will be treated with moderate intensity exercises). Eligible participants attended three session per week. Overnight fast, resting metabolic rate and blood pressure will be assessed. An oral glucose test will be assessed and baseline blood samples will be used for lipoprotein analysis. Pacer test and step test performed in the each session. A regular follow-up visits to department and a final assessment will be made at the end of last week by using questionnaire and resulting improvement will shown in results after completion. Data will be analyzed on SPSS 25.

DETAILED DESCRIPTION:
The study will be a Randomized clinical trial and will be conducted in services hospital lahore. The study will be completed within the duration of ten months. Non probability convenient sampling study technique will be used to collect the data. The sample size of 50 patients will be taken in this study to find the effects of high intensity interval training versus moderate intensity exercises on physical health and cardiorespiratory fitness in obese women.

Patients will be divided into two groups (Group A will be treated with high intensity interval training and Group B will be treated with moderate intensity exercises). Eligible participants attended three session per week. Overnight fast, resting metabolic rate and blood pressure will be assessed. An oral glucose test will be assessed and baseline blood samples will be used for lipoprotein analysis. Pacer test and step test performed in the each session. A regular follow-up visits to department and a final assessment will be made at the end of last week by using questionnaire and resulting improvement will shown in results after completion. Data will be analyzed on SPSS 25.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 17-30 years

  * BMI 25-35kg/m2.
  * Sedentary (< 30 minutes of structured activity per week)
  * Normal glucose tolerance ( fasting glucose <100mg/dL)
  * No use of medications known to affect body composition or metabolism
  * All participants will be non smoker
  * No MI history
  * No previous surgery.
  * Free from known injury or known clinical conditio

Exclusion Criteria:

* BMI < 30 kg/m2 Known clinical condition including family history of sudden death, uncontrolled hypertension, type 1 and type 2 diabetes and cardiovascular diesease. • Participants will be excluded if they report in competitive exericise

Ages: 17 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-02-20 (Estimated)

PRIMARY OUTCOMES:
Step test | 4weeks
  the step test is designed to measured a person's aerobic fitness. Participants steps up and down, on and off, an aerobics- type step for three minutes to increase heart rate and to evaluate the heart's recovery rate during the minute immediately following the step test exercise.
Glucose tolerance test | 4weeks
  The glucose tolerance test is a medical test in which glucose is given and blood samples taken afterward to determine how quickly it is cleared from the blood. The test is usually used to test for diabetes, insulin resistance. an oral glucose tolerance test (OGTT), a standard dose of glucose is ingested by mouth and blood levels are checked two hours later.
Lipoprotein blood test: | 4weeks
  lipoprotein test measures the level of lipoprotein in your blood. Lipoproteins are substances made of protein and fat that carry cholesterol through your bloodstream. Lipoprotein (a) is a type of LDL (bad) cholesterol. A high level of lipoprotein
  (a) may mean you are at risk for heart disease.

CONTACTS AND LOCATIONS:
Overall Officials: madiha younas, MS, Principal Investigator — riphah internationl university
Locations (1):
- Ittefaq Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No